CLINICAL TRIAL: NCT06700291
Title: Preoperative Frailty and Postoperative Neurocognitive Disorders in Geriatric Patients in Georgia
Acronym: FRAILCOG-GE
Status: Recruiting | Type: Observational
Sponsor: New Hospitals Georgia (Other)
Responsible Party: Principal Investigator, Tamar Macharadze, Principle Investigator Dr.Tamar Macharadze, New Hospitals Georgia
Other Study IDs: 01/01
Record Dates: First submitted 2024-11-01; First posted 2024-11-21 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2024-11

CONDITIONS: Frailty
Keywords: Delirium,; Perioperative neurocognitive disorder; Geriatric anaesthesia; Dementia; Frailty
MeSH Terms: conditions — Frailty; Delirium; Dementia | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Surgery — Patient undergoing Anesthesia and Surgery

SUMMARY:
The number of elderly people in the global population is growing, presenting an increasing challenge. Technological advances in medicine have made it possible to perform complex surgeries on geriatric patients, improving the viability of this age group. However, postoperative neurocognitive disorders represent the most common postoperative complications in this demographic, leading to increased morbidity and mortality, a reduced quality of life, and a heightened risk of dementia.

In high-income countries, studies have shown that preoperative frailty is associated with a cascade of postoperative disorders, including cognitive decline, delirium, dementia, and mortality. These complications negatively impact the community as a whole, healthcare staff and services, and the daily lives of those affected and their families. Perioperative neurocognitive disorders are linked to longer hospital stays, increased economic costs, reduced ability to work, and adverse consequences for family members and caregivers.

Frailty is a syndrome characterized by decreased reserve and resistance to stressors, resulting from cumulative declines in multiple physiological systems over time. This leaves individuals less capable of mounting a satisfactory response to stressful events. Frailty is most prevalent in the aging population, with its prevalence increasing exponentially with age.

This study will be the first to investigate preoperative frailty and its association with postoperative cognitive disorders in Georgia. Currently, there is limited information regarding the geriatric population in Georgia. The study will explore the prevalence of preoperative frailty and its impact on postoperative outcomes, including depression, dementia, cognitive dysfunction, delirium, and mortality at 30 days, three months, and one year following anesthesia and surgery.

This pioneering research will provide valuable insights into these disorders in low- and middle-income countries. It will fill a significant gap in the international literature by contributing essential knowledge that is currently lacking in this field.

DETAILED DESCRIPTION:
Investigators will conduct a prospective, observational cohort study to determine the prevalence of frailty in the geriatric population of Georgia, focusing on men and women aged 65 years and older undergoing elective orthopedic surgery. All participants will provide written, informed consent to participate in the study.

Frailty will be assessed using the frail scale test preoperatively, at discharge, three months, and one year postoperatively. Baseline cognitive function will be evaluated using the Montreal Cognitive Assessment (MoCA) and modified Telephone Interview for Cognitive Status (TICSm) test and will enable cognitive screening and the detection of pre-existing cognitive disorders. Postoperative neurocognitive disorders (NCDs) will also be assessed with TICSm at one months, three months, and one year postoperatively through telephone follow-ups.

Delirium will be evaluated preoperatively and twice daily during the patient's hospital stay using the Three-Minute Diagnostic Interview for Confusion Assessment (3D-CAM). If patients require intensive care postoperatively, the Confusion Assessment Method for the ICU (ICU CAM) will also be administered twice daily.

Depression will be measured with the Geriatric Depression Scale (GDS) preoperatively and postoperatively at discharge, and again at one month, three months, and one year. Anxiety will be assessed using a visual analogue scale at baseline, discharge, one month, three months, and one year. The Trail Making Test A and B will be administered preoperatively and at discharge. Pain levels will be measured during each assessment using the Numerical Rating Scale (NRS).

Disability and the ability to perform daily living activities will be evaluated at baseline, three months, and one year postoperatively using the WHO Disability Assessment Schedule (WHODAS.2.0) and Activities of Daily Living -Prevention Instrument test (ADL-PI).

Additionally, investigators will collect demographic and clinical information, including education level, comorbidities, alcohol use, lifestyle factors, and body mass index (BMI). Laboratory tests will also be conducted to explore potential mechanisms underlying postoperative neurocognitive disorders (PND), such as albumin, HbA1c, triglycerides, electrolytes, creatinine, Vitamin D, and interleukin-6 (IL-6).

All assessments and tests originally in English will be translated into Georgian and validated for the Georgian population before being administered to patients in the hospital.

ELIGIBILITY:
Inclusion Criteria:

Male or female patients aged 65 years or older

Scheduled for elective orthopedic surgery (hip or knee arthroplasty with endoprosthesis)

Able to provide informed consent

Exclusion Criteria:

Diagnosis of dementia (any type)

Major psychiatric disorder (e.g., schizophrenia, bipolar disorder, severe depression)

Surgery performed within the past 6 months

Inability to complete neuropsychological assessment due to sensory or communication impairment (e.g., severe vision loss, hearing impairment, language barrier, aphasia)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Male or female patients aged 65y or more, scheduled for elective orthopedic surgery with knee or hip endoprosthesis.
Sampling Method: Probability Sample
Enrollment: 230 (Estimated)
Dates: Start 2023-04-26 (Actual); Primary Completion 2026-04-09 (Estimated); Study Completion 2026-04-09 (Estimated)

PRIMARY OUTCOMES:
Determine the prevalence of preoperative frailty | Frailty assessments will be conducted at baseline preoperatively, on the day of hospital discharge (dependes how many days the patient stay in the hospital), and during follow-up at 3 months and 12 months post-surgery.
  Frailty will be assessed using the FRAIL scale in patients aged 65 years and older undergoing planned orthopedic surgery and will be conducted at four time points: preoperatively, on the day of discharge, and at 3 and 12 months postoperatively.

SECONDARY OUTCOMES:
Correlation between preoperative frailty and postoperative disorders (postoperative delirium, delayed neurocognitive recovery and postoperative neurocognitive disorder) up to one year after surgery . | Frailty: preop, within 12h prior to hospital discharge, and 3 & 12 mo postop; TMT A/B: baseline, within 12h prior to discharge; TICSm: 1, 3 & 12 mo postop; 3D-CAM & ICU-CAM: twice daily from postop day 1 until within 12 hours prior to discharge.
  Frailty will be assessed using the FRAIL scale in patients aged 65 year and older undergoing planned orthopedic surgery. Postoperative delirium,delayed neurocognitive recovery and postoperative neurocognitive disorders will be assessed by following tests: 3D CAM, ICU CAM, Trial Making test A and B, TICSm.
Preoperative demographics and risk factors, including but not limited to age, level of education, and comorbidities, and their correlation with any perioperative neurocognitive disorders up to twelve months following surgery. | Demographic information and risk factors will be collected on baseline.Postopereative outcomes will be collected on the day of discharge from the hospital,1 months, 3 months and 1 year after the surgery.
  Preoperative demographic information and risk factors-including, but not limited to, age, education, and comorbidities-will be collected. Upon study completion, these factors will be analyzed for their correlation with postoperative outcomes
Prevalence of preoperative cognitive impairment | MoCA and TICSm - preoperative;
  Preoperative cognitive impairment will be assessed using both the Montreal Cognitive Assessment (MoCA) and the modified Telephone Interview for Cognitive Status (TICSm).
Correlation between preoperative cognitive impairment and postoperative disorders (postoperative delirium, delayed neurocognitive recovery and postoperative neurocognitive disorder) up to one year after surgery | MoCA and TICSm - preop; TICSm-1,3 and 12 mo postop. 3D-CAM: twice daily from postop day 1 until within 12h prior to hospital discharge; ICU-CAM: twice daily while in ICU; TMT A/B: preop baseline and within 12h prior to discharge regardless of stay length
  Preoperative cognitive impairment will be assessed using both the Montreal Cognitive Assessment (MoCA) and the modified Telephone Interview for Cognitive Status (TICSm). Postoperative delirium,delayed neurocognitive recovery and postoperative neurocognitive disorders will be assessed by following tests: 3D CAM, ICU CAM, Trial Making test A and B, TICSm.
Determine the prevalence of depression in older adults presenting for anesthesia and surgery. | Assessment time points: preoperative baseline
  Depression will be assessed using the Geriatric Depression Scale (GDS) preoperatively.
Preoperative depression in older adults in Georgia presenting for anesthesia and surgery correlation with postoperative depression during different time points | Baseline, on the day of discharge, one months and three months postop,one year after the surgery
  Depression will be essessed with geriatric depression scale teset preoperatively, on the day of discharge , one months and three months postop and one year after surgery.
To determine the mortality rate up to one year after anesthesia and surgery | In hospital,1 months, 3 months and 12 months postoperatively.
  Mortality will be recorded through hospital records and follow-up telephone contact with the a family member at one months, three months and twelve months after surgery.
Patient disability change among older adults in Georgia from the preoperative to postoperative period using WHO Disability Assessment Schedule 2.0 | WHODAS 2. questionary will be used Preoperatively, 3 months and 12 months postoperatively.
  Disability will be assessed using the WHO Disability Assessment Schedule 2.0 (WHODAS 2.0) questionaries. They will be administered peroperatively, 3 months and 12 months postoperatively. Acording the scores these assessments will help to evaluate changes in functional status over time.Allowing anylysis of the impact of surgery and anesthesia on patients disability .
Patient quality of life change among older adults in Georgia from the preoperative to postoperative period using Daily Living prevention instrument questionary. | Daily Living prevention instrument questionaries will be used Preoperatively, 3 months and 12 months postoperatively.
  Patient quality of life will be assessed using the Daily Living prevention instrument questionaries. They will be administered peroperatively, 3 months and 12 months postoperatively. According the scores these assessments will help to evaluate changes in daily living over time.Allowing anylysis of the impact of surgery and anesthesia on patients functional ability .

CONTACTS AND LOCATIONS:
Overall Officials: Tamar Macharadze, Dr, Principal Investigator — David Tvildiani Medical University
Locations (1):
- New Hospitals, Tbilisi, Georgia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Darsalia T, Evered L, Macharadze T. Preoperative frailty and postoperative neurocognitive disorders in older adults in Georgia: study protocol for a prospective, observational cohort study. BMJ Open. 2025 Oct 20;15(10):e101245. doi: 10.1136/bmjopen-2025-101245. PMID 41120173